CLINICAL TRIAL: NCT02177669
Title: Test-Retest Variability of Quick Contrast Sensitivity Function Testing
Status: Completed | Type: Observational
Sponsor: Nova Southeastern University (Other)
Collaborators: Adaptive Sensory Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 05291468Exp; R21EY023720 (NIH); Adaptive Sensory Technology (Other Grant/Funding Number: Adaptive Sensory Technology)
Record Dates: First submitted 2014-06-26; First posted 2014-06-30 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Healthy
Keywords: Normal, healthy individuals without ocular disease; Ages 20-89; English speaking; Visual acuity better than 20/25

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Normals without ocular disease
  Interventions: Other: quick Contrast Sensitivity Function test

INTERVENTIONS:
Other: quick Contrast Sensitivity Function test

SUMMARY:
The contrast sensitivity function (CSF) provides a comprehensive characterization of spatial vision and predicts functional vision better than visual acuity, but long testing times prevent its psychophysical assessment in clinical applications. Dr. Luis Lesmes et al. (2010) developed the qCSF method to obtain precise CSF measurements in only 30-50 trials using a computerized software program that presents letters on a large monitor that are identified by a patient similar to typical visual acuity testing with an eye chart. The quick CSF method is a Bayesian adaptive method that estimates the full shape of the CSF, and the test duration is only about 3-6 minutes. Some preliminary testing has been performed at other sites with this test in patients with vision loss due to amblyopia and glaucoma, but data from individuals without eye disease who have normal visual acuity has not been systematically collected with the latest version of this test procedure across a wide range of ages. In addition, we aim to gain a better understanding of the typical test-retest variability that is obtained between-sessions that are about a week apart from individuals with good ocular health and visual acuity.

ELIGIBILITY:
Inclusion Criteria:

* Ages 20-89
* Normal distance visual acuity in each of both eyes (20/20)
* Absence of ocular disease
* Able and willing to complete contrast sensitivity testing
* Provide informed consent

Exclusion Criteria:

* Any ocular disease
* Refractive errors >6D
* Inability to understand study or communicate responses (cognitive impairment)
* Unable to understand, read and speak English fluently

Ages: 20 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals between the ages of 20-89 without ocular disease will be recruited from among patients seen in the Primary Eye Care Clinic at the Nova Southeastern University's The Eye Care Institute in Davie-Ft. Lauderdale, FL, as well as faculty, students and staff at this institution.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-06; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
95% coefficient of repeatability across subjects | test-retest at 2 visits about a week apart
  We will evaluate various contrast sensitivity metrics that are generated by the computer program: (i) AULCSF or area under the curve for the log contrast sensitivity function (CSF), (ii) CSF acuity or the cutoff-frequency at which sensitivity=2.0 is calculated, and (iii) contrast sensitivity at various spatial frequencies (i.e. 1.5, 3, 6, 12, 18.5 cycles per degree), obtained with testing performed binocularly, with the better eye monocularly, and with the better eye using a NoIR 4% transmission filter. Within subject, the data will be analyzed as differences between the two values obtained at the two sessions, which can then be used to determine a 95% coefficient of repeatability across subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Ava K Bittner, OD, PhD, Principal Investigator — Nova Southeastern University; College of Optometry
Locations (1):
- Nova Southeastern University; College of Optometry, Fort Lauderdale, Florida, United States

REFERENCES:
- [Background] Dorr M, Lesmes LA, Lu ZL, Bex PJ. Rapid and reliable assessment of the contrast sensitivity function on an iPad. Invest Ophthalmol Vis Sci. 2013 Nov 5;54(12):7266-73. doi: 10.1167/iovs.13-11743. PMID 24114545
- [Background] Lesmes LA, Lu ZL, Baek J, Albright TD. Bayesian adaptive estimation of the contrast sensitivity function: the quick CSF method. J Vis. 2010 Mar 30;10(3):17.1-21. doi: 10.1167/10.3.17. PMID 20377294